CLINICAL TRIAL: NCT01904903
Title: SAFE-HEaRt: A Pilot Study Assessing the Cardiac SAFEty of HER2 Targeted Therapy in Patients With HER2 Positive Breast Cancer and Reduced Left Ventricular Function
Brief Title: Cardiac Safety Study in Patients With HER2 + Breast Cancer
Acronym: SAFE-HEaRt
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML 28685
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: HER2 Positive Breast Cancer; Left Ventricular Function Systolic Dysfunction
Keywords: Breast Cancer HER2 Positive; Cardiac Safety
MeSH Terms: interventions — Trastuzumab; pertuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HER2 therapies, cardiac medications (Other): Cardiac intervention - beta-blockers and ACE-inhibitors titrated to the maximum tolerated doses
  Oncology intervention - patients will receive one of the three following HER2 targeted therapies at the discretion of the treating oncologist:
  * Trastuzumab: loading dose of 8 mg/kg IV, followed by a maintenance dose of 6 mg/kg every 3 weeks, or a loading dose of 4 mg/kg followed by a maintenance dose of 2 mg/kg every week.
  * Pertuzumab: loading dose of 840 mg IV, followed by 420 mg IV every 3 weeks, administered concomitantly with trastuzumab.
  * Ado trastuzumab emtansine (TDM1): 3.6mg/kg IV every three weeks.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Ado Trastuzumab Emtansine

INTERVENTIONS:
Drug: Trastuzumab — HER2 therapy
  Other Names: Herceptin
Drug: Pertuzumab — HER2 therapy
  Other Names: Perjeta
Drug: Ado Trastuzumab Emtansine — HER2 therapy
  Other Names: Kadcyla

SUMMARY:
HER2 positive breast cancer cells have more HER2 receptor (a protein on the surface of cells) than normal breast cells. Approximately 30% of patients with breast cancer have HER2 positive breast cancer. Before HER2 targeted therapies (i.e. treatments that directly block the receptor HER2) were developed, patients with HER2 positive breast cancer had a very aggressive form of disease. With the use of trastuzumab, an anticancer drug that directly targets the receptor HER2, and more recently, pertuzumab and ado-trastuzumab emtansine, patients are able to live longer and have better control of their cancer.

Unfortunately the use of HER2 targeted therapies can increase the risk of heart problems and for this reason these treatments were only studied and approved for patients with normal heart function.

In this study we plan to give HER2 targeted therapies to patients with HER2 positive breast cancer and mildly decreased heart function along with concomitant evaluation by a heart doctor (called cardiologist) and appropriate medications to strengthen the heart. We will do frequent monitoring of the heart function with a test called echocardiogram that will give us a detailed "picture" of the heart. We will also draw blood along with routine blood tests to try to understand why some patients develop heart problems and others do not. The study will take a maximum of 12 months and patients will be monitored for 6 additional months.

We hypothesize that it is safe to administer HER2 targeted therapies to patients with breast cancer and mildly decreased heart function, i.e. LVEF between 40 and 50%, while on appropriate heart medications.

DETAILED DESCRIPTION:
Title: A pilot study evaluating the cardiac safety of HER2 targeted therapy (non-lapatinib) in patients with HER2 positive breast cancer and reduced left ventricular function Phase: Pilot study Study Duration: 4 years with up to 5 additional years of follow up Study Center(s): 3 centers will be participating: MedStar Washington Hospital Center (MWHC), MedStar Georgetown University Hospital (MGUH) and Memorial Sloan Kettering Cancer Center (MSKCC) Primary Objective: To evaluate the cardiac safety of HER2 targeted therapy (non-lapatinib) in patients with HER2 positive breast cancer and reduced left ventricular ejection fraction (LVEF) when given concomitantly with cardiac treatment.

Secondary Objectives:

* To evaluate time to development of cardiac event or asymptomatic worsening of cardiac function
* Absolute changes in LVEF
* Delays in HER2 therapy attributed to cardiac causes
* Correlations between echocardiographic myocardial strain
* cTnI and hs-cTnT at baseline and over time with cardiac events and asymptomatic worsening of cardiac function Sample size: 30 patients

Diagnosis and Main Inclusion Criteria:

* HER2 positive breast cancer, stage I-IV.
* Mildly decreased cardiac function (LVEF between 40 and 49%) prior to or while receiving non-lapatinib HER2 targeted therapy

Cardiac Intervention:

- Beta-blockers and ACE-inhibitors titrated to the maximum tolerated doses

Oncology study Products, Doses, Routes, Regimens:

* Trastuzumab: loading dose of 8 mg/kg IV, followed by a maintenance dose of 6 mg/kg every 3 weeks, or a loading dose of 4 mg/kg followed by a maintenance dose of 2 mg/kg every week.
* Pertuzumab: loading dose of 840 mg IV, followed by 420 mg IV every 3 weeks, administered concomitantly with trastuzumab.
* Ado-trastuzumab emtansine: 3.6mg/kg IV every three weeks. Note: both trastuzumab and pertuzumab may be administered alone or in combination with other systemic or radiation therapy.

Duration of drug administration: Maximum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient diagnosed with stage I-IV breast cancer
* HER2 positive breast cancer, defined by immunohistochemical staining for HER2 protein of 3+ intensity and/or amplification of the HER2 gene on fluorescence in situ hybridization (FISH) ≥ 2.0 on breast specimen or biopsy of a metastatic site
* LVEF < 50% and ≥ 40% documented in echocardiogram done within the last 30 days
* HER2 therapy naïve or currently receiving non-lapatinib HER2 targeted therapy
* Patient receiving or planning to receive trastuzumab, trastuzumab with pertuzumab or ado-trastuzumab emtansine, for at least 3 months, alone or in combination with other systemic treatment or radiation
* Age ≥ 18 years
* Patient is willing and able to comply with protocol required assessments and procedures

Exclusion Criteria:

* Previous hospitalization due to documented heart failure in the last 12 months
* Current signs or symptoms of heart failure or ischemia
* History of arrhythmia requiring pharmacological or electrical treatment
* Concomitant use of anthracyclines or use of anthracyclines in the last 50 days
* Pregnant or lactating patients. Patients of childbearing potential must implement contraceptive measures during study treatment and for 7 months after last dose of treatment drug and must have negative urine or serum pregnancy test within 7 days prior to registration.
* History of significant neurologic or psychiatric disorders including psychotic disorders or dementia that would prohibit the understanding and giving of informed consent.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Swain, MD, Principal Investigator — Washington Cancer Institute at MedStar Washington Hospital Center
Locations (2):
- United States (2):
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia

REFERENCES:
- [Result] Lynce F, Barac A, Geng X, Dang C, Yu AF, Smith KL, Gallagher C, Pohlmann PR, Nunes R, Herbolsheimer P, Warren R, Srichai MB, Hofmeyer M, Cunningham A, Timothee P, Asch FM, Shajahan-Haq A, Tan MT, Isaacs C, Swain SM. Prospective evaluation of the cardiac safety of HER2-targeted therapies in patients with HER2-positive breast cancer and compromised heart function: the SAFE-HEaRt study. Breast Cancer Res Treat. 2019 Jun;175(3):595-603. doi: 10.1007/s10549-019-05191-2. Epub 2019 Mar 9. PMID 30852761
- [Result] Lynce F, Barac A, Tan MT, Asch FM, Smith KL, Dang C, Isaacs C, Swain SM. SAFE-HEaRt: Rationale and Design of a Pilot Study Investigating Cardiac Safety of HER2 Targeted Therapy in Patients with HER2-Positive Breast Cancer and Reduced Left Ventricular Function. Oncologist. 2017 May;22(5):518-525. doi: 10.1634/theoncologist.2016-0412. Epub 2017 Mar 17. PMID 28314836

RESULTS

PARTICIPANT FLOW:
Groups:
- HER2 Therapies, Cardiac Medications: Cardiac intervention - beta-blockers and ACE-inhibitors titrated to the maximum tolerated doses
  Oncology intervention - patients will receive one of the three following HER2 targeted therapies at the discretion of the treating oncologist:
  * Trastuzumab: loading dose of 8 mg/kg IV, followed by a maintenance dose of 6 mg/kg every 3 weeks, or a loading dose of 4 mg/kg followed by a maintenance dose of 2 mg/kg every week.
  * Pertuzumab: loading dose of 840 mg IV, followed by 420 mg IV every 3 weeks, administered concomitantly with trastuzumab.
  * Ado trastuzumab emtansine (TDM1): 3.6mg/kg IV every three weeks.
  Trastuzumab: HER2 therapy
  Pertuzumab: HER2 therapy
  Ado Trastuzumab Emtansine: HER2 therapy
Period: Overall Study
Arm/Group | HER2 Therapies, Cardiac Medications
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | HER2 Therapies, Cardiac Medications
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Latino Black | 17
  Non-Latino White | 12
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Complete Planned Oncologic Therapy Without the Development of a Cardiac Event or Asymptomatic Worsening of Cardiac Function.
Description: Cardiac events are defined as any of the following:
  * Presence of symptoms attributable to heart failure as confirmed by a cardiologist
  * Cardiac arrhythmia requiring pharmacological or electrical treatment
  * Myocardial infarction
  * Sudden cardiac death or death due to myocardial infarct, arrhythmia or heart failure
  Asymptomatic worsening of cardiac function defined as:
  - Asymptomatic decline in LVEF > 10% points from baseline and/or EF < 35% corroborated by a confirmatory echocardiogram in 2-4 weeks
  Planned oncologic therapy is defined as:
  * In the adjuvant setting: completion of 1 year total of HER2 targeted therapy. If a patient already received part of the planned HER2 targeted therapy prior to enrollment in this trial, planned oncologic therapy will be achieved when a total of 1 year is completed.
  * In the metastatic setting: cessation of treating regimen due to progressive disease or non-cardiac toxicity or non-cardiac death.
Time Frame: Up to 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | HER2 Therapies, Cardiac Medications
Number analyzed (Participants) | 30
Participants | 27

2. Secondary Outcome: Median Time to Development of an Event Defined as Cardiac Event or Asymptomatic Worsening of Left Ventricular Dysfunction, Among Patients Who Developed One Event.
Time Frame: Up to 18 months.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | HER2 Therapies, Cardiac Medications
Number analyzed (Participants) | 30
days | 220 [201 to 252.5]

3. Secondary Outcome: Absolute Changes in LVEF During HER2 Targeted Therapy Between Baseline and End of Treatment
Description: Difference in LVEF between end of treatment and baseline
Time Frame: Up to 18 months.
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | HER2 Therapies, Cardiac Medications
Number analyzed (Participants) | 30
percent ejection fraction | 4.21 (3.4)

4. Secondary Outcome: HER2 Therapy Holds Attributed to Proportion of Patients With Symptomatic or Asymptomatic Cardiotoxicity.
Description: Proportion of patients that had a hold because of symptomatic or asymptomatic cardiotoxicity.
  Hold is defined as any delay or discontinuation of HER2 targeted therapy due to cardiac toxicity. One cycle of HER2 targeted therapy will be considered 3 weeks. One therapy hold will be defined as any 3-week HER2 targeted therapy missed dose or 1/3 if one weekly trastuzumab dose. For patients who had a hold and resumed HER2 targeted therapy, duration of treatment hold will be described.
Time Frame: Up to 12 months.
Measure: Number; unit: proportion of participants
Arm/Group | HER2 Therapies, Cardiac Medications
Number analyzed (Participants) | 30
proportion of participants | 0.1

5. Secondary Outcome: Correlation of Global Longitudinal Myocardial Strain With Cardiac Events and Asymptomatic Worsening of Cardiac Function
Time Frame: Up to 18 months.
Population: There were too few clinical events to assess correlations
Arm/Group | HER2 Therapies, Cardiac Medications
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation of Standard Cardiac Troponin I and Highly Sensitive Cardiac Troponin T With Cardiac Events and Asymptomatic Worsening of Cardiac Function
Time Frame: Up to 18 months.
Population: This outcome was not analyzed. There were too few clinical events to assess correlations.
Arm/Group | HER2 Therapies, Cardiac Medications
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HER2 Therapies, Cardiac Medications
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HER2 Therapies, Cardiac Medications (N=30)
Cardiac event (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT01904903/Prot_SAP_000.pdf